CLINICAL TRIAL: NCT01391039
Title: Microbubble Contrast Ultrasound and Transient Elastography Imaging of Early Breast Cancer
Brief Title: Diagnostic Study of Early Breast Cancer Using Ultrasound
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RJ07062011
Record Dates: First submitted 2011-06-15; First posted 2011-07-11 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Ductal Carcinoma In-situ
Keywords: Ductal Carcinoma In-situ; Contrast Ultrasound; Microinvasion; Elastography
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast perfusion and elastography arm (Experimental): Intravenous injection of microbubble contrast agent and elastography
  Interventions: Drug: Perflutren lipid microsphere

INTERVENTIONS:
Drug: Perflutren lipid microsphere — Intravenous injection of 10 microL/kg once prior to ultrasound examination
  Other Names: Definity

SUMMARY:
This is a pilot study designed to investigate new techniques to guide the appropriate diagnosis and treatment of Ductal Carcinoma In-situ (DCIS). The microvascularity and stiffness of the lesion may be prognostic factors that can guide the need for more or less extensive therapy or perhaps only imaging follow-up may be needed.

DETAILED DESCRIPTION:
Women who have imaging findings suggestive of DCIS, who are having breast ultrasound and who are candidates for surgery will be eligible. They will receive a contrast-enhanced breast ultrasound after the intravenous injection of a microbubble contrast agent which will show the microvascularity. A subset of women will also have ultrasound elastography performed of the abnormality to evaluate its stiffness.

ELIGIBILITY:
Inclusion Criteria:

* A woman with imaging signs suggesting a diagnosis of DCIS who is scheduled for ultrasound and a biopsy is eligible for the study.
* At least 18 years of age

Exclusion Criteria:

* Pregnant or possibly pregnant or breast feeding
* Unable to provide informed consent
* Drug or multiple allergies
* Known cardiac shunts
* Known cardiac or chronic pulmonary disease
* Hypersensitivity to perflutren

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Evidence of the presence of angiogenic tumour vasculature in patients diagnosed with DCIS utilizing contrast enhanced ultrasound. | The participant will be followed up till the results of the biopsy, an expected average of 3 months.

SECONDARY OUTCOMES:
Measurement of transient shear wave elastography . | The participant will be followed up till the results of the biopsy, an expected average of 3 months.
  The quantitative intralesional measurement of shear wave modulus will be compared to the angiogenesis imaging and biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta A Jong, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada